CLINICAL TRIAL: NCT02734706
Title: Efficacy of a Supplement Capsule Containing LRC™ (L. Reuteri NCIMB 30242) on Managing Cholesterol Levels in Adults
Brief Title: Efficacy of a LRC™ (L. Reuteri NCIMB 30242) Capsule on Managing Cholesterol in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UAS Labs LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15LCHU
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LRC™ capsule (Experimental)
  Interventions: Dietary Supplement: LRC™ capsule
- Placebo capsule (Placebo Comparator)
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Dietary Supplement: LRC™ capsule — Twice per day (BID), 9 weeks
  Arms: LRC™ capsule
Other: Placebo capsule — Twice per day (BID), 9 weeks
  Arms: Placebo capsule

SUMMARY:
To investigate the effect of a supplement capsule containing LRC™ (L. reuteri NCIMB 30242), taken twice daily with lunch and dinner (NLT 2.5E9 CFU per dose), versus placebo capsule on serum low density lipoprotein (LDL)-cholesterol in otherwise healthy hypercholesterolemic adults after 9 weeks of product consumption.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 20 to 75 years.
* LDL-C ≥ 3.40 mmol/L at visits V0 and V2-1 (<15% variation between visits V0 and V2-1).
* TG < 4.00 mmol/L (checked at visits V0 and V2-1).
* BMI between 23.0 to 32.5 kg/m2.
* Subject understands and accepts to follow the dietary recommendations advisable for hypercholesterolemic patients (according to NCEP-ATP III guidelines)
* Judged by the investigators as compliant (>80%) with product consumption (check at V2-1), and motivated.
* Subjects taking stable doses of thyroid hormone and anti-hypertensive agents will be permitted, as long as these are continued equivalently throughout the duration of study.
* Agreement to maintain current level of physical activity throughout the study.
* If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System); Intrauterine devices; Vasectomy of partner.
* Voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Use of cholesterol lowering prescription drugs within the last 6 months.
* Use of plant sterols, omega 3, fish oil, soy protein, soluble oat fiber, psyllium seed husk, or other cholesterol lowering non-prescription supplements within last 1 month.
* History of chronic use of alcohol (>2 drinks/d).
* History of heavy smoking (≥20 cigarettes/d).
* Use of systemic antibodies, corticosteroids, androgens, or phenytoin.
* Immune-compromised subjects (e.g. AIDS, lymphoma, subjects undergoing long-term corticosteroid treatment).
* Subject having experienced any cardiovascular event (myocardial infarction, coronary artery bypass, or other major surgical procedures) in the last 6 months.
* Subjects with elevated LDL-C (≥ 3.40 mmol/L) and high (>20%) CVD risk estimated by the Framingham risk score.
* Previously diagnosed Type I or Type II diabetes or any other endocrine disorders such as adrenal insufficiency, Cushing's disease, hyperthyroidism, hypopituitarism or polycystic ovary syndrome.
* Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters.
* Subject currently involved in a clinical trial or in an exclusion period following participation in another clinical trial.
* History of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year).
* Clinically significant abnormal laboratory results at screening.
* Chronic user of probiotics or fibre laxative (greater than 2 doses/wk), or stimulant laxatives.
* History of eating disorders.
* Exercise greater than 15 miles/wk or 4,000 kcal/wk.
* For female subjects: Pregnancy, breast feeding, or intent to get pregnant.
* Allergy or sensitivity to test product ingredients.
* Allergy or sensitivity to all 3 antibiotics (Clindamycin, Erythromycin and Ampicillin).
* Diagnosis of anemia or bleeding disorders

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-03; Primary Completion 2018-11 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Serum LDL-cholesterol after 9 weeks of product consumption. | 9 weeks

SECONDARY OUTCOMES:
Serum LDL-cholesterol after 6 weeks of product consumption. | 6 weeks
Serum total cholesterol after 6 and 9 weeks of product consumption. | 6 and 9 weeks
Serum HDL-cholesterol after 6 and 9 weeks of product consumption. | 6 and 9 weeks
Serum non-HDL-cholesterol after 6 and 9 weeks of product consumption. | 6 and 9 weeks
Serum triglycerides after 6 and 9 weeks of product consumption. | 6 and 9 weeks
Serum apolipoprotein B-100 after 6 and 9 weeks of product consumption. | 6 and 9 weeks
Serum hs-CRP after 9 weeks of product consumption. | 9 weeks
Plasma fibrinogen after 9 weeks of product consumption. | 9 weeks
Plasma homocysteine after 9 weeks of product consumption. | 9 weeks
GI health questionnaire score after 6 and 9 weeks of product consumption. | 6 and 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada